CLINICAL TRIAL: NCT04759664
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of Topically Administered LUT014 in Metastatic Colorectal Cancer Patients With EGFR Inhibitor Induced Acneiform Lesions
Brief Title: LUT014 for the Reduction of Dose-Limiting Acneiform Lesions Associated With EGFRI Treatment of mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lutris Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L-02-01
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: EGFRI Induced Acneiform Lesions
Keywords: EGFRI, Acneiform, Acneiform lesions, Acneiform rash, EGFRI induced skin toxicities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LUT014 Gel (Dose 1) (Experimental)
  Interventions: Drug: LUT014 Gel (Dose 1)
- LUT014 Gel (Dose 2) (Experimental)
  Interventions: Drug: LUT014 Gel (Dose 2)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LUT014 Gel (Dose 1) — Topical gel
  Arms: LUT014 Gel (Dose 1)
Drug: LUT014 Gel (Dose 2) — Topical gel
  Arms: LUT014 Gel (Dose 2)
Drug: Placebo — LUT014 matching placebo topical gel
  Arms: Placebo

SUMMARY:
The study evaluates the efficacy and safety of two strengths of LUT014 Gel topically applied once a day for 4 weeks, compared to placebo, in metastatic colorectal cancer (mCRC) patients who developed Grade 2 or non-infected Grade 3 EGFRI induced acneiform lesions

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with mCRC;
2. Currently being treated with an FDA approved monoclonal antibody EGFRI for the treatment of mCRC, including but not limited to Erbitux® (cetuximab) Injection and Vectibix® (panitumumab) Injection, as directed by the approved labeling;
3. Grade 2 or Grade 3 non-infected acneiform lesions at the Screening and Baseline;
4. A reversed score of no more than 44 for the skin-specific questions (first 13 questions) of the FACT-EGFRI-18 HRQoL questionnaire at the Screening and Baseline;
5. Age ≥18 years at the time of signing the informed consent form (ICF);
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2;
7. Expected life expectancy greater than 3 months;
8. Subject can understand and sign the ICF, can communicate with the Investigator, can understand and comply with the requirements of the protocol, and can apply the study drug by himself/herself or has a care giver that can apply the drug;
9. Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 0);

Exclusion Criteria:

1. Active infection within the treatment area or in other body areas that requires initiation of systemic antibiotics ;
2. Significant skin disease other than EGFRI induced acneiform lesions within the same body areas planned for study drug application;
3. Has a beard that would interfere with administration of study drug and assessment of study endpoints (scoring of lesions);
4. Any cancer other than mCRC within 3 years of Screening, except for carcinoma in situ of the cervix;
5. Any condition which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study;
6. Clinically relevant serious co-morbid medical conditions including, but not limited to, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, active central nervous system (CNS) disease uncontrolled by standard of care, known positive status for human immunodeficiency virus (HIV) and/or active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements;
7. Pregnant or lactating;
8. Treatment with an EGFRI other than the FDA approved monoclonal antibody EGFRI for the treatment of mCRC within 30 days or 5 half-lives of the drug prior to Screening, whichever is longer;
9. Treatment with a serine/threonine-protein kinase B-Raf (B-Raf) inhibitor, including but not limited to Zelboraf® (vemurafenib), Tafinlar® (dabrafenib), Braftovi® (encorafenib), and Nexavar® (sorafenib), within 30 days or 5 half-lives of the drug prior to Screening, whichever is longer. Patients whose mCRC is being treated with a monoclonal antibody EGFRI in combination with a B-Raf inhibitor, such as Erbitux® (cetuximab) Injection in combination with Braftovi® (encorafenib) Capsules, will not be eligible to participate in this trial;
10. Treatment with a systemic corticosteroid 14 days prior to Baseline or treatment with a topical corticosteroid to the face, neck, or upper portion of the anterior or posterior chest within 7 days prior to Baseline (Day 0). Patients receiving systemic corticosteroids for 24 hours or less only at the time of chemotherapy infusions (for the prevention or treatment of chemotherapy-induced nausea and vomiting) will be allowed to enroll into this study;
11. Treatment with a topical antibiotic to the face, neck, or upper portion of the anterior or posterior chest within 7 days prior to Baseline (Day 0);
12. Initiation of treatment with systemic antibiotic(s) < 28 days prior to Baseline (Day 0) or any change in dose or frequency of systemic antibiotic(s) within 28 days prior to Baseline. Patients that undergo a washout from systemic antibiotic(s) will be allowed to participate in this trial as long as no systemic antibiotics are taken within 7 days prior to Baseline and they meet all other eligibility criteria;
13. Treatment with any other topical medication applied to the face, neck, or upper portion of the anterior or posterior chest within 7 days prior to Baseline (Day 0).
14. Treatment with an oral retinoid within 30 days or 5 half-lives of the drug prior to Baseline (Day 0), whichever is longer. Patients that undergo a washout from oral retinoids will be allowed to participate
15. Treatment with another investigational drug within 30 days or 5 half-lives of drug prior to Screening, whichever is longer;
16. Known hypersensitivity to the inactive ingredients of the study drug (active or placebo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects in each treatment group who reached treatment success | Four weeks (28 days)
  Treatment success will be defined as an improvement (decrease) of at least one grade in the severity of the acneiform lesions from baseline to Day 28, based on CTCAE V5.0 skin and subcutaneous tissue disorders grading scale OR an improvement (increase) of at least 5 points in the total score for the skin-specific (first 13 questions) of the FACT-EGFRI-18 HRQoL questionnaire, from baseline to Day 28, with the exception of subjects who:
  1. their dose of EGFRI was decreased, delayed, or stopped during the RDPBC treatment period
  2. initiated treatment with topical or systemic antibiotic(s) for the treatment of their acneiform lesions during the RDPBC treatment period
  3. experience an increase in the dose or frequency of the systemic antibiotic(s) relative to Baseline during the RDPBC treatment period
  4. are discontinued from study drug (active or placebo) during the RDBPC treatment period due to worsening of their acneiform lesions

SECONDARY OUTCOMES:
Change in the severity of acneiform lesions based on CTCAE grading scale from baseline to Days 7, 14, 21, 28, and 55. For subjects enrolled in the OLE, the change from pre-dose Day 28 to Days 35, 42, 49, 56, and 84 will also be evaluated; | 8-16 weeks (56-84 days)
Change in the FACT-EGFRI-18 questionnaire total score for the skin-specific questions from baseline to Days 7, 14, 21, 28, and 55. For subjects enrolled in the OLE, the change from pre-dose Day 28 to Days 35, 42, 49, 56, and 84 will also be evaluated; | 8 -16 weeks (56-84 days)
Relative change in the FACT-EGFRI-18 HRQoL questionnaire | 8 weeks (56 days)
  Relative change in the FACT-EGFRI-18 score for the skin-specific questions from D0 to D7,14,21,28, 55 compared to the maximal possible improvement in the score from D0; and the relative change from D28 to D35,42,49,56,84 compared to the maximal possible improvement in the score from D28 for OLE subjects.
Proportion of subjects whose dose of EGFRI was decreased, delayed, or stopped during the RDPBC and the OLE treatment period | 4 weeks (28 days)
Number of AEs and the number and percentage of subjects with AEs | 8 weeks (6 days)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Innovative Clinical Research Institute, Glendale, California
  - UCLA, Santa Monica, California
  - Miami Dermatology & Laser Research, Miami, Florida
  - Miami Dermatology and Laser Institute, Miami, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Appalachian Regional Healthcare, Hazard, Kentucky
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack Meridian Health, Neptune City, New Jersey
  - Memorial Sloane Kettering, New York, New York
  - New York Cancer and Blood Specialists, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center Investigational Drug Service, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Israel (3):
  - Assuta Ashdod, Ashdod
  - E. Wolfson Medical Center, Holon
  - Shaara Zedek Medical Center, Jerusalem